CLINICAL TRIAL: NCT03217851
Title: Prevalence Survey of Plasmodium Falciparum Antimalarial Drug Resistance Markers in Greater Mekong Subregion
Brief Title: Prevalence Survey of Antimalarial Drug Resistance Markers
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Worldwide Antimalarial Resistance Network (Network); Mahidol Oxford Tropical Medicine Research Unit (Other); Myanmar Oxford Clinical Research Unit (Other); Shoklo Malaria Research Unit (Other); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other); Oxford University Clinical Research Unit, Vietnam (Other); Cambodia Oxford Medical Research Unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: BAKMAL 1701
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-05

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Prevalence Survey; Antimalarial Drug
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Blood Specimen Collection; Dried Blood Spot Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Collect blood for malaria diagnostic testing (blood smear and/or rapid diagnostic test) and dried blood spot on filter paper
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Presenting P. falciparum Malaria
  Interventions: Diagnostic Test: Blood Collection; Diagnostic Test: Dried Blood Spot

INTERVENTIONS:
Diagnostic Test: Blood Collection — blood smear and/or rapid diagnostic
Diagnostic Test: Dried Blood Spot — Dried Blood Spot on filter paper

SUMMARY:
Study is cross-sectional and observational with one-time dried-blood spot sample collection from persons with laboratory-confirmed uncomplicated Plasmodium falciparum malaria (mixed or monoinfection). Samples will be analysed for the presence of molecular markers of resistance to ACT partner drugs (gene amplifications and/or other mutations in pfmdr1, gene amplifications of pfpm2, and additional mutations which may be identified during the course of the trial) in the first instance. Testing to detect additional markers of antimalarial drug resistance will also be performed where feasible. Prevalence of mutations will be summarized and mapped to provide intelligence on antimalarial drug resistance in the region of interest.

DETAILED DESCRIPTION:
Malaria Malaria is caused by a mosquito-borne, protozoan parasite belonging to the genus Plasmodium. Of the five species of Plasmodium that infect humans, Plasmodium falciparum is the most deadly and is responsible for the majority of malaria disease and death. Every year, falciparum malaria causes disease in hundreds of millions of people living in the tropics and subtropics, killing a million or more according to some estimates. The vast majority of these deaths occur in sub-Saharan Africa, mostly among young children and infants. When treated with effective antimalarial drugs, malaria can be cured completely.

Antimalarial drug resistance The emergence in Southeast Asia and the subsequent global spread of drug resistant malaria was a major factor contributing to the failure of the first global malaria eradication campaign in the mid-20th century (1). The widespread implementation of highly effective artemisinin-based combination therapy (ACT) for malaria has contributed to significant gains in global control and elimination efforts and has brought malaria eradication back on the agenda, 40 years after the first global malaria eradication campaign was abandoned (2). However the gains seen in the past decade are now at risk as parasite resistance to artemisinin compounds has been confirmed in Southeast Asia and threatens Africa once again (3-8). In the absence of effective vaccines, it is critical to prolong the usable life of antimalarial drugs by judicious implementation of treatment strategies.

Primary Objective To measure prevalence of established and candidate molecular markers of drug resistant malaria in Greater Mekong Subregion

Secondary Objective To map the geographical and temporal changes in prevalence of molecular markers of antimalarial drug resistance in Greater Mekong Subregion

Funder: EXPERTISE FRANCE Grant reference number: Expertise France reference 15SANIN211

ELIGIBILITY:
Inclusion Criteria:

* Patients (6 months - 75 years) with confirmed uncomplicated P. falciparum infection
* Written informed consent obtained (by parents/guardian in case of children less than 18 years old)

Exclusion Criteria:

Patients presenting signs of severe malaria* will be excluded from the survey to prevent any delay in the management of the patient.

*Guideline for the treatment of Malaria-3rd edition, WHO (27) Severe falciparum malaria is defined as one or more of the following, occurring in the absence of an identified alternative cause and in the presence of P.falciparum asexual parasitaemia.

* Impaired consciousness: A Glasgow comma score < 11 in adults or Blantyre coma score < 3 in children
* Prostration: Generalized weakness so that the person is unable to sit, stand or walk without assistance.
* Multiple convulsions: More than two episodes within 24 h
* Acidosis: A base deficit of > 8 mEq/L or, if not available a plasma bicarbonate level of < 15 mmol/L or venous plasma lactate ≥ 5 mmol/L. Severe acidosis manifests clinically as respiratory distress (rapid, deep, laboured breathing).
* Hypoglycaemia: Blood or plasma glucose < 2.2 mmol/L (<40 mg/dL)
* Severe malarial anaemia: Haemoglobin concentration ≤ 5 g/dL or a haematocrit of ≤ 15% in children < 12 years of age (< 7 g/dL and < 20%, respectively, in adults) with a parasite count > 10,000/µL
* Renal impairment: Plasma or serum creatinine > 265 µmol/L (3 mg/dL) or blood urea > 20 mmol/L
* Jaundice: Plasma or serum bilirubin > 50 µmol/L (3 mg/dL) with a parasite count > 100,000/ µL
* Pulmonary oedema: Radiologically confirmed or oxygen saturation < 92% on room air with a respiratory rate > 30/min, often with chest indrawing and crepitations on auscultation
* Significant bleeding: Including recurrent or prolonged bleeding from the nose, gums or venepuncture site; haematemesis or melaena
* Shock: Compensated shock is defined as capillary refill ≥ 3 s or temperature gradient on leg (mid to proximal limb), but no hypotension. Decompensated shock is defined as systolic blood pressure < 70 mm Hg in children or < 80 mm Hg in adults, with evidence of impaired perfusion (cool peripheries or prolonged capillary refill)
* Hyperparasitaemia: P.falciparum parasitaemia > 10%

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients age 6 months - 75 years presenting at study site with confirmed P. falciparum infection
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Prevalence and geospatial trends of molecular markers, information to assist definition of treatment policies | 3 years

SECONDARY OUTCOMES:
Visualization and dissemination of molecular marker prevalence data to inform public health officials, researchers, policymakers and key stakeholders | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, Prof, Study Director — Shoklo Malaria Research Unit; Frank Smithuis, Prof, Study Director — Myanmar Oxford Clinical Research Unit; Mayfong Mayxay, Prof, Principal Investigator — Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit; Nguyen Thanh Thuy Nhien, Dr, Principal Investigator — Oxford University Clinical Research Unit, Vietnam; Arjen M. Dondorp, PhD, Principal Investigator — Mahidol Oxford Clinical Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.wwarn.org/working-together/sharing-data/data-usage